CLINICAL TRIAL: NCT04271709
Title: The Manhattan Vision Screening and Follow-Up Study (NYC-SIGHT)
Brief Title: Manhattan Vision Screening and Follow-Up Study (NYC-SIGHT)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Lisa Hark, PhD, MBA, Professor of Ophthalmic Sciences, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: AAAR9162; U01DP006436 (NIH)
Record Dates: First submitted 2020-02-13; First posted 2020-02-17 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Glaucoma; Vision Impairment and Blindness; Cataract; Diabetic Retinopathy; Eye Diseases
Keywords: Vision Screening; Follow-up Eye Care; Vulnerable Populations; New York City
MeSH Terms: conditions — Glaucoma; Vision Disorders; Blindness; Cataract; Diabetic Retinopathy; Eye Diseases

STUDY DESIGN:
Intervention Model Description: 2:1 randomization by housing development
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Intervention (Active Comparator): Consented subjects living in buildings randomized to the Patient Navigator Intervention arm who failed the screening and needed vision correction received free eyeglasses, which were fitted by an optician at the housing building. If they were referred to an ophthalmologist for a follow-up eye exam, they received enhanced support with patient navigators to assist with follow-up eye exams at Columbia Ophthalmology or Harlem Hospital, specifically eye exam appointment scheduling and arranging transportation over a 1-year period.
  Interventions: Behavioral: Enhanced Intervention Using Patient Navigators
- Usual Care (Placebo Comparator): Consented subjects living in buildings randomized to Usual Care arm who failed the screening and needed vision correction were given an eyeglasses prescription and a list of optical shops within 1 mile from their home. These subjects who are referred to an ophthalmologist for a follow-up eye exam were only scheduled for their initial appointment at either Columbia Ophthalmology or Harlem Hospital. They did not receive enhanced support. Scheduling this initial appointment allowed tracking of adherence.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Enhanced Intervention Using Patient Navigators — Enhanced support by patient navigators assisted with follow-up eye exam appointment scheduling and arranging transportation over a 1-year period.
  Arms: Enhanced Intervention
Other: Usual Care — Usual Care subjects who failed the screening and needed vision correction were given an eyeglasses prescription and a list of optical shops within 1 mile from their home. These subjects did not receive enhanced support. Scheduling this initial appointment will allow tracking of adherence.
  Arms: Usual Care

SUMMARY:
The investigators are conducting a 5-year prospective, 2:1 cluster-randomized controlled trial, funded by the Centers for Disease Control (CDC), which provides vision screenings to underserved New York City residents living in affordable housing buildings in Harlem and Washington Heights.

DETAILED DESCRIPTION:
This study aims to increase engagement, detection and management of glaucoma, vision impairment, cataracts, and other eye diseases in vulnerable populations living in New York City. This study considers disparities by race, ethnicity, gender, geography, and socioeconomic status using innovative approaches such as patient navigators. Individuals over the age of 40 living in New York City Housing Authority (NYCHA) Housing buildings are eligible.

ELIGIBILITY:
Inclusion Criteria:

* Individuals over age 40
* Living independently in NYCHA housing building or attending DFTA Senior Center
* Willing to answer COVID-19 symptom questions
* Willing to consent for 2 vision screening visits at baseline and 12-month follow-up

Exclusion Criteria:

* Self-reported terminal illness with life expectancy less than 1 year
* Inability to provide informed consent due to dementia or other reasons

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 749 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2025-09-29 (Actual); Study Completion 2026-09-29 (Estimated)

PRIMARY OUTCOMES:
Proportion of Subjects with Visual Acuity Worse than 20/40 | 2 years
  Visual acuity (VA) is a measure of the spatial resolution of the visual processing system. Visual acuity will be measured in each eye and measured as ≤20/40 or >20/40. Since there are two best corrected distance visual acuity measurements per person (right eye and left eye), the visual acuity in the worse eye will be used in the analysis and reported at the patient level, rather than the eye level. Visual acuity analysis will be handled as a dichotomous variable and the proportion of subjects with visual acuity 20/40 or worse will be considered abnormal.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa A. Hark, PhD, RD, Principal Investigator — Columbia University
Locations (1):
- Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sapru S, Berktold J, Crews JE, Katz LJ, Hark L, Girkin CA, Owsley C, Francis B, Saaddine JB. Applying RE-AIM to evaluate two community-based programs designed to improve access to eye care for those at high-risk for glaucoma. Eval Program Plann. 2017 Dec;65:40-46. doi: 10.1016/j.evalprogplan.2017.06.006. Epub 2017 Jun 21. PMID 28689028
- [Background] Hark L, Acito M, Adeghate J, Henderer J, Okudolo J, Malik K, Molineaux J, Eburuoh R, Zhan T, Katz LJ. Philadelphia Telemedicine Glaucoma Detection and Follow-up Study: Ocular Findings at Two Health Centers. J Health Care Poor Underserved. 2018;29(4):1400-1415. doi: 10.1353/hpu.2018.0103. PMID 30449754
- [Background] Pizzi LT, Waisbourd M, Hark L, Sembhi H, Lee P, Crews JE, Saaddine JB, Steele D, Katz LJ. Costs of a community-based glaucoma detection programme: analysis of the Philadelphia Glaucoma Detection and Treatment Project. Br J Ophthalmol. 2018 Feb;102(2):225-232. doi: 10.1136/bjophthalmol-2016-310078. Epub 2017 Jun 27. PMID 28655730
- [Background] Waisbourd M, Shafa A, Delvadia R, Sembhi H, Molineaux J, Henderer J, Pizzi LT, Myers JS, Hark LA, Katz LJ. Bilateral Same-day Laser Peripheral Iridotomy in the Philadelphia Glaucoma Detection and Treatment Project. J Glaucoma. 2016 Oct;25(10):e821-e825. doi: 10.1097/IJG.0000000000000409. PMID 26950579
- [Background] Hark LA, Radakrishnan A, Madhava M, Anderson-Quinones C, Fudemberg S, Robinson D, Myers JS, Zhan T, Adeghate J, Hegarty S, Leite S, Leiby BE, Stempel S, Katz LJ. Awareness of ocular diagnosis, transportation means, and barriers to ophthalmology follow-up in the Philadelphia Telemedicine Glaucoma Detection and Follow-up Study. Soc Work Health Care. 2019 Aug;58(7):651-664. doi: 10.1080/00981389.2019.1614711. Epub 2019 May 23. PMID 31120381
- [Background] Hark LA, Adeghate J, Katz LJ, Ulas M, Waisbourd M, Maity A, Zhan T, Hegarty S, Leiby BE, Pasquale LR, Leite S, Saaddine JB, Haller JA, Myers JS. Philadelphia Telemedicine Glaucoma Detection and Follow-Up Study: Cataract Classifications Following Eye Screening. Telemed J E Health. 2020 Aug;26(8):992-1000. doi: 10.1089/tmj.2019.0170. Epub 2019 Nov 13. PMID 31721654
- [Background] Adeghate JO, Hark LA, Brown H, Henderer JD, Waisbourd M, Molineaux J, Malik K, Maity A, Chuang D, Donches K, Heres C, Eburuoh R, Schardt M, Yu D, Ramsey F, Myers JS, Katz LJ. Philadelphia glaucoma detection and treatment project: ocular outcomes and adherence to follow-up at a single health centre. Can J Ophthalmol. 2019 Dec;54(6):717-722. doi: 10.1016/j.jcjo.2019.03.003. Epub 2019 Sep 19. PMID 31836105
- [Background] Hark LA, Myers JS, Pasquale LR, Razeghinejad MR, Maity A, Zhan T, Hegarty SE, Leiby BE, Waisbourd M, Burns C, Divers M, Molineaux J, Henderer JD, Haller JA, Katz LJ. Philadelphia Telemedicine Glaucoma Detection and Follow-up Study: Intraocular Pressure Measurements Found in a Population at High Risk for Glaucoma. J Glaucoma. 2019 Apr;28(4):294-301. doi: 10.1097/IJG.0000000000001207. PMID 30946709
- [Background] Hark LA, Myers JS, Ines A, Jiang A, Rahmatnejad K, Zhan T, Leiby BE, Hegarty S, Fudemberg SJ, Mantravadi AV, Waisbourd M, Henderer JD, Burns C, Divers M, Molineaux J, Pizzi LT, Murchison AP, Saaddine J, Pasquale LR, Haller JA, Katz LJ. Philadelphia Telemedicine Glaucoma Detection and Follow-up Study: confirmation between eye screening and comprehensive eye examination diagnoses. Br J Ophthalmol. 2019 Dec;103(12):1820-1826. doi: 10.1136/bjophthalmol-2018-313451. Epub 2019 Feb 15. PMID 30770354
- [Background] Hark LA, Katz LJ, Myers JS, Waisbourd M, Johnson D, Pizzi LT, Leiby BE, Fudemberg SJ, Mantravadi AV, Henderer JD, Zhan T, Molineaux J, Doyle V, Divers M, Burns C, Murchison AP, Reber S, Resende A, Bui TDV, Lee J, Crews JE, Saaddine JB, Lee PP, Pasquale LR, Haller JA. Philadelphia Telemedicine Glaucoma Detection and Follow-up Study: Methods and Screening Results. Am J Ophthalmol. 2017 Sep;181:114-124. doi: 10.1016/j.ajo.2017.06.024. Epub 2017 Jun 30. PMID 28673747
- [Background] Leiby BE, Hegarty SE, Zhan T, Myers JS, Katz LJ, Haller JA, Waisbourd M, Burns C, Divers M, Molineaux J, Henderer J, Brodowski C, Hark LA. A Randomized Trial to Improve Adherence to Follow-up Eye Examinations Among People With Glaucoma. Prev Chronic Dis. 2021 May 20;18:E52. doi: 10.5888/pcd18.200567. PMID 34014814
- [Background] Newman-Casey PA, Hark LA, Rhodes LA. It Is Time to Rethink Adult Glaucoma Screening Recommendations. J Glaucoma. 2023 Feb 1;32(2):69-71. doi: 10.1097/IJG.0000000000002146. Epub 2022 Nov 25. No abstract available. PMID 36696354
- [Result] De Moraes CG, Hark LA, Saaddine J. Screening and Interventions for Glaucoma and Eye Health Through Telemedicine (SIGHT) Studies. J Glaucoma. 2021 May 1;30(5):369-370. doi: 10.1097/IJG.0000000000001782. No abstract available. PMID 33428354
- [Result] Hark LA, Kresch YS, De Moraes CG, Horowitz JD, Park L, Auran JD, Gorroochurn P, Stempel S, Maruri SC, Stidham EM, Banks AZ, Saaddine JB, Lambert BC, Pizzi LT, Sapru S, Price S, Williams OA, Cioffi GA, Liebmann JM. Manhattan Vision Screening and Follow-up Study in Vulnerable Populations (NYC-SIGHT): Design and Methodology. J Glaucoma. 2021 May 1;30(5):388-394. doi: 10.1097/IJG.0000000000001795. PMID 33492894
- [Result] Hark LA, Lin WV, Hirji S, Gorroochurn P, Horowitz JD, Diamond DF, Park L, Wang Q, Auran JD, Maruri SC, Henriquez DR, Sharma T, Valenzuela I, Liebmann JM, Cioffi GA, Friedman DS, Harizman N. Manhattan Vision Screening and Follow-Up Study (NYC-SIGHT): Subanalysis of Referral to Ophthalmology. Curr Eye Res. 2024 Feb;49(2):197-206. doi: 10.1080/02713683.2023.2269614. Epub 2024 Jan 18. PMID 37812506
- [Result] Horowitz JD, Adeghate JO, Karani R, Henriquez DR, Gorroochurn P, Sharma T, Park L, Wang Q, Diamond DF, Harizman N, Auran JD, Maruri SC, Liebmann JM, Cioffi GA, Hark LA. Manhattan Vision Screening and Follow-Up Study: (NYC-SIGHT)Tele-Retinal Image Findings and Importance of Photography. Telemed J E Health. 2024 Mar;30(3):664-676. doi: 10.1089/tmj.2023.0134. Epub 2023 Sep 1. PMID 37651209
- [Result] Hark LA, Tan CS, Kresch YS, De Moraes CG, Horowitz JD, Park L, Auran JD, Gorroochurn P, Stempel S, Maruri SC, Besagar S, Saaddine JB, Lambert BC, Pizzi LT, Sapru S, Price S, Williams OA, Cioffi GA, Liebmann JM. Manhattan Vision Screening and Follow-Up Study in Vulnerable Populations: 1-Month Feasibility Results. Curr Eye Res. 2021 Oct;46(10):1597-1604. doi: 10.1080/02713683.2021.1905000. Epub 2021 Apr 19. PMID 33726583
- [Result] Hark LA, Horowitz JD, Gorroochurn P, Park L, Wang Q, Diamond DF, Harizman N, Auran JD, Maruri SC, Henriquez DR, Carrion J, Muhire RSM, Kresch YS, Pizzi LT, Jutkowitz E, Sapru S, Sharma T, De Moraes CG, Friedman DS, Liebmann JM, Cioffi GA. Manhattan Vision Screening and Follow-up Study (NYC-SIGHT): Baseline Results and Costs of a Cluster-Randomized Trial. Am J Ophthalmol. 2023 Jul;251:12-23. doi: 10.1016/j.ajo.2023.01.019. Epub 2023 Jan 21. PMID 36690289
- [Result] Sapru S, Price SM, Hark LA, Rhodes LA, Newman-Casey PA. Recruiting Populations at Higher Risk for Glaucoma and Other Eye Diseases Experiencing Eye Health Disparities. Ophthalmic Epidemiol. 2024 Jun;31(3):220-228. doi: 10.1080/09286586.2023.2232038. Epub 2023 Jul 5. PMID 37408319
- [Result] Hark LA, Wang Y, Gorroochurn P, Simon PR, Maruri SC, Henriquez DR, Diamond DF, Horowitz JD, Park L, Wang Q, Auran JD, Carrion J, Friedman DS, Liebmann JL, Cioffi GA, Harizman N. Manhattan Vision Screening and Follow-up Study (NYC-SIGHT): a nested cross-sectional assessment of falls risk within a cluster randomised trial. Br J Ophthalmol. 2024 Nov 22;108(12):1761-1768. doi: 10.1136/bjo-2022-323052. PMID 38609163
- [Result] Hark LA, Gorroochurn P, Tang H, Torres DR, Blackburn B, Maruri SC, Diamond DF, Harizman N, Wang Q, Wang Y, Liebmann JM, Cioffi GA, Horowitz JD, Park L. Improvement in vision-related quality-of-life using the NEI-VFQ-9 over 1-year in the Manhattan Vision Screening and Follow-up Study (NYC-SIGHT). Graefes Arch Clin Exp Ophthalmol. 2025 Jul;263(7):2069-2079. doi: 10.1007/s00417-024-06727-z. Epub 2025 Jan 15. PMID 39812799
- [Result] Wang Q, Valenzuela IA, Harizman N, Gorroochurn P, Torres DR, Maruri SC, Diamond DF, Horowitz JD, Friedman DS, De Moraes CG, Cioffi GA, Liebmann JM, Hark LA. Glaucoma Screening and Referral Risk Factors in a High-Risk Population: Follow-Up Study of the Manhattan Vision Screening Study. J Glaucoma. 2025 Mar 1;34(3):164-174. doi: 10.1097/IJG.0000000000002521. Epub 2024 Nov 26. PMID 39792808
- [Result] Diamond DF, Kresch YS, Gorroochurn P, Park L, Horowitz JD, Wang Q, Maruri SC, Henriquez DR, Harizman N, Carrion J, Liebmann JM, Cioffi GA, Hark LA. Manhattan Vision Screening and Follow-up Study (NYC-SIGHT): Vision and refractive error results. Clin Exp Optom. 2025 Mar;108(2):183-190. doi: 10.1080/08164622.2024.2322523. Epub 2024 Mar 7. PMID 38452798
- [Result] Hark LA, Gorroochurn P, Pizzi LT, Jutkowitz E, Goulak AM, Maruri SC, Harizman N, Horowitz JD, Park L, Wang Q, Diamond DF, Valenzuela IA, Torres DR, Wang Y, Sharma T, Liebmann JM, Cioffi GA. Patient Navigators Improve In-Office Eye Exam Adherence After Community Eye Screenings in a Randomized Clinical Trial: NYC-SIGHT Study. Am J Ophthalmol. 2025 Jun;274:54-66. doi: 10.1016/j.ajo.2025.02.030. Epub 2025 Feb 26. PMID 40015588
- [Derived] Diamond DF, Hirji S, Xing SX, Gorroochurn P, Horowitz JD, Wang Q, Park L, Harizman N, Maruri SC, Henriquez DR, Liebmann JM, Cioffi GA, Hark LA. Manhattan Vision Screening and Follow-Up Study (NYC-SIGHT): optometric exam improves access and utilization of eye care services. Graefes Arch Clin Exp Ophthalmol. 2024 May;262(5):1619-1631. doi: 10.1007/s00417-023-06344-2. Epub 2024 Jan 8. PMID 38189973